CLINICAL TRIAL: NCT03335917
Title: Oxygen Transport in Normobaric vs. Hypobaric Hypoxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 0209-17-FB
Record Dates: First submitted 2017-09-05; First posted 2017-11-08 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Hypoxia, Altitude; Exercise
MeSH Terms: conditions — Altitude Sickness; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized,Counter Balanced, Repeated Measures, Crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normobaric Normoxia (Placebo Comparator): This will serve as the exercise only control trial
  Interventions: Other: Exercise
- Normobaric Hypoxia (Experimental): This arm will provide hypoxia by reducing the amount of oxygen concentration without changing the barometric pressure
  Interventions: Other: Hypoxia; Other: Exercise
- Hypobaric Hypoxia (Experimental): This arm will provide hypoxia by reducing the barometric pressure without changing the oxygen concentration (terrestrial altitude exposure)
  Interventions: Other: Hypoxia; Other: Exercise

INTERVENTIONS:
Other: Hypoxia — Participants will be exposed to hypoxia by reducing barometric pressure or by reducing oxygen concentration
  Arms: Hypobaric Hypoxia; Normobaric Hypoxia
Other: Exercise — Graded cycling exercise to volitional fatigue

SUMMARY:
1) Oxygen Transport in Normobaric versus Hypobaric Hypoxia. 2) The purpose of this study is to examine acute responses in arterial and muscle tissue oxygenation during incremental exercise in normobaric versus hypobaric hypoxia. 3) The participants in this study will consist of 12 recreationally active males and females between the ages of 19 and 45.Recreationally active is defined as participating in moderate to vigorous physical activity for 30 minutes at least 3 days per week.4) Subjects will complete an incremental cycle test to volitional fatigue in three conditions in a randomized counter-balanced order, normobaric normoxia (20.9% O2, 730 mmHg), normobaric hypoxia (14.3% O2, 730 mmHg) and hypobaric hypoxia (20.9% O2, 530mmHg). Two of the three trials will be conducted in an environmental chamber to simulate normobaric normoxia at 350 m (elevation of Omaha, NE) and normobaric hypoxia at 3094 m (elevation of Leadville, CO). The hypobaric hypoxia trial will be conducted in Leadville, Colorado at 3094 m. Trials will be separated by at least two days. Rating of perceived exertion, heart rate, blood oxygenation, respiration rate, muscle tissue oxygenation, and whole body gases will be analyzed during the trials. 5) There is no follow-up as a part of this study.

DETAILED DESCRIPTION:
The specific objective of the study is to identify physiological differences between acute exposure to normobaric and hypobaric hypoxia.

The majority of well controlled research investigating the physiological effects of altitude have been conducted in chambers that create a hypoxic environment by reducing the fraction of oxygen in the environment (normobaric hypoxia). With actual altitude exposure, the fraction of oxygen remains constant but the barometric pressure providing the driving force for the binding of oxygen to hemoglobin is reduced (hypobaric hypoxia). Both circumstances should in theory lead to the same partial pressure of oxygen. Recent research has called the normobaric hypoxia model for altitude exposure into question and demonstrates that normobaric and hypobaric hypoxia may lead to differential physiological responses. Indeed, research from our lab has shown a higher heart rate and lower arterial oxygen saturation with hypobaric hypoxia compared to normobaric hypoxia. Others have also documented a further decrease in physical performance lower ventilatory response and pH, and higher oxidative stress in hypobaric hypoxia compared to normobaric hypoxia. The ability to interchange these methods of achieving a hypoxic environment is not without controversy. our lab has recently investigated the skeletal muscle transcriptional response after exposure to both normobaric and hypobaric hypoxia. The investigators found only limited differences in the muscle transcriptional response between the two forms of hypoxia despite differences in arterial oxygen saturation and heart rate. Clearly, more work is needed to determine the physiological aspects that may be differentially affected by normobaric and hypobaric hypoxia. This project will fill the knowledge gap of differences between forms of hypoxia in the resting and exercise response. Specifically, we will non-invasively determine the muscle oxygenation (NIRS) response that may help explain the lack of difference between the forms of hypoxia on the muscle transcriptional response. Furthermore, while heart rate has been shown to be differentially affected, no data currently exists on the variability of heart rate. It will determine the effects on heart rate variability (a marker of autonomic nervous system function and strong predictor of mortality). The addition of this data to the body of literature will have an impact on the physiological understanding of the effects of hypoxia and have major implications to the interpretation of previous research based on the experimental model used.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be recreationally active Recreationally active is defined as participating in moderate to vigorous physical activity for 30 minutes at least 3 days per week.-females or males between the ages of 19 and 45.
* All participants must be considered "low risk" according to ACSM risk stratification.
* participants must be free from any ECG or blood pressure abnormalities as assessed during maximal testing.

Exclusion Criteria:

* All subjects who are considered higher than "low risk" according to the ACSM risk stratification guidelines will be excluded from this study.
* Any participant under 19 years of age or over the age 45 and who list any health related condition that may interfere or become exacerbated by participating in this research would be excluded from this study.
* Participants taking any prescription drugs, other than female contraceptives, will be excluded from participation.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Change in Muscle Oxygenation | change from baseline at 0 minutes after exercise
  % O2 sat in muscle using NIRS

CONTACTS AND LOCATIONS:
Overall Officials: Dustin R Slivka, PhD, Principal Investigator — University of Montana
Locations (1):
- University of Nebraska at Omaha, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
No plan to make IPD available to other researchers.